CLINICAL TRIAL: NCT01578564
Title: Phase I, Open-label, Dose Escalation Study to Assess Safety and Tolerability of SOR-C13 in Subjects With Advanced Solid Tumors Commonly Known to Express the TRPV6 Ion Channel
Brief Title: Safety and Tolerability Study of SOR-C13 in Subjects With Advanced Cancers Commonly Known to Express the TRPV6 Channel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Soricimed Biopharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOR-C13 01
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Cancer
Keywords: Cancer; Ovarian Cancer; TRPV6 Calcium channel
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms | interventions — SOR-C13

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SOR-C13 (Experimental)
  Interventions: Drug: SOR-C13

INTERVENTIONS:
Drug: SOR-C13 — Intravenous solution for infusion, potential dose range 1.375 mg/kg to 6.12 mg/kg, dosing frequency 2 cycles with a cycle consisting of infusions on days 1-3 and days 8-10 followed by a 11 day off period

SUMMARY:
The purpose of this study is to determine the safety and tolerability of the drug SOR-C13 when given as an intravenous infusion in patients with ovarian cancer or other cancers known to over express the TRPV6 calcium channel.

ELIGIBILITY:
Inclusion criteria

* Males and females ≥ 18 years of age
* Subjects with a histologic diagnosis of solid tumor cancers of epithelial origin.
* Subjects with advanced refractory cancer for which standard curative or palliative measures do not exist or are no longer effective. There is no limitation on the number or types of prior therapy.
* Subjects must have recovered from major infections and/or surgical procedures and, in the opinion of the investigator, not have a significant active concurrent medical illness precluding protocol treatment.
* ECOG (Eastern Cooperative Oncology Group) Performance Score ≤ 1.
* Life expectancy of greater than 12 weeks.
* Subjects must have adequate organ and marrow function as defined below:

  1. hemoglobin ≥9.0 g/dL (≥5.6 mmol/L)
  2. white blood cells ≥3,000/mm³(≥3×10⁹/L)
  3. absolute neutrophil count ≥1,500/mm³ (≥1.5×10⁹/L)
  4. platelets ≥100,000/μL (≥100×10⁹/L)
  5. total bilirubin ≤1.5× upper limit of normal(ULN)
  6. AST/ALT/AP ≤2.5× ULN (ALT/AST ≤5.0x ULN in case of documented liver metastases
  7. creatinine ≤1.5× ULN
  8. albumin ≥3.0 g/dL (≥30 g/L)
  9. INR ≤1.4
* Ability to understand and voluntarily sign the informed consent document

Exclusion Criteria:

* Chemotherapy, immunotherapy, radiotherapy, biologic or any investigational therapy will not be allowed within either 30 days, or 5 half lives (whichever is longer) prior to study drug administration.
* History or clinical evidence of central nervous system (CNS) tumor involvement (metastases) or other known clinically relevant CNS pathology (e.g., epilepsy, seizure, paresis, aphasia, cerebellar disease, severe brain injury, psychosis).
* Concurrent malignancy other than the solid tumor under investigation, requiring active treatment.
* History of clinically significant allergic reaction attributed to any injected compound.
* History of any of the following cardiovascular events or conditions within the past 6 months prior to enrolment: myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, New York Heart Association Class ≥ II chronic heart failure, hypokalemia, significant arrhythmia*; QTc interval >430 msec or use of drugs that prolong the QT interval at screening; family history of long QT syndrome.(* Significant arrhythmias are defined as symptoms of syncope or severe palpitations (palpitations requiring referral to cardiac monitoring), or ECG findings of supraventricular tachycardia (including ventricular fibrillation) or ventricular ectopy (ventricular premature depolarization).
* Clinically significant and uncontrolled major medical condition(s) that places the subject at an unacceptably high risk for toxicities. These include, but are not limited to: active infections, symptomatic pulmonary disease, inadequate pulmonary function, seizure disorder, psychiatric illness.
* Current use of more than one antihypertensive medication.
* For patients receiving antihypertensive medication:systolic blood pressure < 120 mmHg and/or diastolic blood pressure < 70 mmHg at screening.
* A known diagnosis of human immunodeficiency virus (HIV) infection or acquired immune deficiency syndrome (AIDS), acute or chronic hepatitis B or hepatitis C infection, as determined by medical history.
* Major surgical procedure within 4 weeks prior to enrolment.
* Lactating or pregnant female.
* Females of childbearing potential and males not using adequate birth control.
* Current treatment or treatment within 4 weeks of screening with bisphosphonates.
* Screening serum calcium levels < 2.20 mmol/L [8.8 mg/dL] (after correction for serum albumin
* History of acute pancreatitis within 12 months prior to screening
* Known hypoparathyroidism, pseudohypoparathyroidism, or vitamin D deficiency, or clinical evidence of other conditions known to associated with hypocalcemia, including:, hypoalbuminemia, hyperphosphatemia, hypomagnesemia
* Current treatment or treatment within 4 weeks of screening with drugs known to reduce serum calcium levels, including: bisphosphonates, antiepileptic drugs, cinacalcet, macrolide antibiotics (such as erythromycin, azithromycin), large doses of corticosteroids (>20 mg/day of prednisone or equivalent), or any IV use of corticosteroids. In addition, long-term use (defined as ongoing use for ≥4 weeks) of corticosteroids within 8 weeks of screening is prohibited
* Any history of a venous thromboembolic event (VTE), including deep vein thrombosis (DVT) or pulmonary embolism (PE)
* Current treatment or treatment within 7 days of screening with a vitamin K antagonist, such as warfarin. Patients who require anticoagulation due to their central line may receive an alternative agent, such as low molecular weight heparin (LMWH).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-07; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Toxicity graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Over 21 days from initial administration

SECONDARY OUTCOMES:
Plasma levels of SOR-C13 | Pre-treatment and up to 4 hours post-treatment on Study Days 1, 3, 8 and 10

CONTACTS AND LOCATIONS:
Overall Officials: Toney T Ilenchuk, MS, PhD, Study Director — Soricimed Biopharma Inc
Locations (3):
- MD Anderson Cancer Center, Houston, Texas, United States
- Canada (2):
  - Juravinski Cancer Center, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario